CLINICAL TRIAL: NCT05058911
Title: Randomized Controlled Trial of Internet-delivered Exposure-based Cognitive Behavior Therapy vs. Internet-delivered Traditional Cognitive Behavior Therapy for Patients With Fibromyalgia
Brief Title: Exposure-based Cognitive Behavior Therapy vs Traditional Cognitive Behavior Therapy for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Maria Hedman-Lagerlöf, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-03302
Record Dates: First submitted 2021-09-08; First posted 2021-09-28 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Fibromyalgia
Keywords: cognitive behavior therapy; randomized controlled trial; internet-delivered treatment
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with repeated measurments and two conditions: the experimental group (Exp-CBT) and an active control group (T-CBT).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered exposure-based cognitive behavior therapy (Exp-CBT) (Experimental): 10-week self-help treatment delivered via a secure online platform, with regular therapist support.
  Interventions: Behavioral: Internet-delivered exposure-based cognitive behavior therapy
- Internet-delivered traditional cognitive behavior therapy (T-CBT) (Active Comparator): 10-week self-help treatment delivered via a secure online platform, with regular therapist support.
  Interventions: Behavioral: Internet-delivered traditional cognitive behavior therapy

INTERVENTIONS:
Behavioral: Internet-delivered exposure-based cognitive behavior therapy — The primary treatment component is exposure to stimuli (situations and activities) that give rise to pain, distress, and unwanted emotional responses. The treatment proceeds in accordance with functional analysis. Exercises are tailored for the patient so that, for example, individuals whose main coping strategy is to be overly active (i.e., persistence behavior) are encouraged to sit down and observe pain and other aversive bodily sensations as they arise. The protocol also includes regular exercises where the participant is encouraged to observe and name physical sensations without acting on them.
  Other Names: Exp-CBT
  Arms: Internet-delivered exposure-based cognitive behavior therapy (Exp-CBT)
Behavioral: Internet-delivered traditional cognitive behavior therapy — This treatment is based on components typical of T-CBT for FM, such as relaxation, activity planning or pacing, cognitive restructuring techniques and stress management strategies.
  Other Names: T-CBT
  Arms: Internet-delivered traditional cognitive behavior therapy (T-CBT)

SUMMARY:
Fibromyalgia (FM) is a common medical condition characterized by chronic generalized musculoskeletal pain, fatigue, and a series of additional somatic and psychiatric problems that give rise to distress, functional impairment, and substantial societal costs. The most extensively evaluated treatment for FM is traditional cognitive behavior therapy (T-CBT) which typically appears to have small to moderate effects when compared to waitlist, attention control, treatment as usual or other active nonpharmacological therapies. Internet-delivered exposure-based cognitive behavior therapy (Exp-CBT) where the patient willingly and systematically engages with stimuli associated with pain and pain-related distress has shown promising controlled effects versus a waiting-list but has never been compared to T-CBT in a randomized controlled trial. In this randomized controlled trial, self-recruited adults with FM (N=260) are randomly assigned (1:1) to 10 weeks of internet-delivered Exp-CBT or internet-delivered T-CBT and complete self-report questionnaires to measure symptoms and therapeutic processes up to 12 months after treatment. Primary outcome is the relative effect of Exp-CBT and T-CBT on FM severity as modelled using linear mixed models fitted on weekly Fibromyalgia Impact Questionnaire sum scores over the treatment period, testing the hypothesis of Exp-CBT superiority based on the coefficient for the time × group interaction. The investigators will also calculate the number of treatment completers in each treatment condition, defined as having commenced module five out of eight treatment modules. Cost-effectiveness and mediational processes are investigated in secondary analyses. The investigators expect this trial to be of notable clinical significance as it will provide valuable information about the value of Exp-CBT in helping patients with FM as compared to using other interventions.

DETAILED DESCRIPTION:
FM is a common problem with substantial negative consequences. The most widely evaluated psychological treatment for FM is T-CBT which usually has small to moderate controlled effects on pain, mood and functional impairment. Based on one pilot study and one wailist-controlled RCT, Exp-CBT appears to have promising effects on FM but this treatment has not yet been compared to an active control condition. The present study aims to compare internet-delivered Exp-CBT to internet-delivered T-CBT in a randomized controlled trial.

Participants in Exp-CBT and T-CBT are encouraged to work with self-help texts and complete regular homework exercises via a secure treatment platform. Both treatments are 10 weeks long, equally exhaustive, and involve approximately the same level of therapist support.

Primary outcome is the relative effect of Exp-CBT and T-CBT on FM severity as modelled using linear mixed models fitted on weekly Fibromyalgia Impact Questionnaire sum scores over the treatment period, testing the hypothesis of Exp-CBT superiority based on the coefficient for the time × group interaction. The investigators will also calculate the number of treatment completers in each treatment condition, defined as having commenced module five out of eight treatment modules. Detailed information regarding analysis of clinical efficacy is provided in the supplementary file.

In addition to clinical efficacy, the investigators will also investigate cost-effectiveness and mediational processes. The primary hypothesis is that Exp-CBT is significantly more efficacious than T-CBT in reducing FM severity, i.e., the Fibromyalgia Impact Questionnaire (FIQ) composite score indicative of symptoms and functional status, from the baseline assessment to the 10-week assessment.

ELIGIBILITY:
Inclusion Criteria:

* Living in Sweden
* Access to the internet
* Completed pre-treatment assessment
* If on psychotropic medication, dose kept stable for at least 4 weeks before randomization and the participant agrees to keep it constant during treatment

Exclusion Criteria:

* Severe depression (≥ 30 on the Montgomery Åsberg Depression Rating Scale-Self Rated [MADRS-S] at screening)
* Suicidal ideation (≥ 4 on the suicide item of the MADRS-S at screening),
* Psychosis
* Alcohol or substance use disorder as primary diagnosis or likely to severely interfere with treatment
* Ongoing psychological treatment
* Pregnancy (>29 wk gestation)
* Another somatic condition that requires immediate treatment and/or is deemed to be the primary condition
* Insufficient knowledge of the Swedish language or insufficient computer skills to benefit from the text-based online treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change in FM severity over the main phase, as modelled using data from all 11 assessments from the pre-treatment assessment, weekly to the primary endpoint (10 weeks). | Screening, Pre-treatment, weekly up to 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  The Fibromyalgia Impact Questionnaire, FIQ. Self-rated, range 0-100. Higher score indicate higher FM severity.

SECONDARY OUTCOMES:
Change in pain over the main phase, as modelled using data from all 11 assessments from the pre-treatment assessment, weekly to the primary endpoint (10 weeks). | Screening, Pre-treatment, weekly up to 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  The Fibromyalgia Impact Questionnaire, FIQ-Pain subscale. Self-rated, range 0 to 10, a higher score indicates more pain.
Change in pain over the main phase, as modelled using data from the pre-treatment assessment and primary endpoint (10 weeks) | Pre-treatment, 10 weeks. Secondary analyses incorporate 6- and 12-MFU assessments.
  Brief Pain Inventory-Short Form, BPI-Sf. Self-rated, range 0-10. A higher score indicates more pain.
Change in fatigue over the main phase, as modelled using data from the pre-treatment assessment and primary endpoint (10 weeks) | Pre-treatment, 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  Fatigue Severity Scale, FSS. Self-rated, range 9-63. A higher score indicates greater fatigue severity
Change in anxiety over the main phase, as modelled using data from the pre-treatment assessment and primary endpoint (10 weeks) | Pre-treatment, 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  GAD-2. Self-rated, range: 0-6. A higher score indicates more general anxiety.
Change in depression over the main phase, as modelled using data from the pre-treatment assessment and primary endpoint (10 weeks) | Pre-treatment, 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  PHQ-2. Self-rated, range: 0-6. A higher score indicates more depressive symptoms.
Change in functional impairment over the main phase, as modelled using data from the pre-treatment assessment and primary endpoint (10 weeks). | Pre-treatment, 10 weeks, Secondary analyses incorporate 6- and 12-months follow-up assessments.
  12-item WHO Disability Assessment Schedule 2.0, WHODAS 2.0. Self-rated, range: 0-100. A higher score indicates more disability.
Change in quality of life over the main phase, as modelled using data from the pre-treatment assessment and primary endpoint (10 weeks). | Pre-treatment, 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  Brunnsviken Brief Quality of Life Inventory, BBQ. Self-rated, range 0 to 96, a higher score indicates better quality of life
Global impression of perceived change at post-treatment | 10 weeks
  Patient Global Impression of Change, PGIC. Self-rated, range no change [or condition has got worse] to a great deal better, and a considerable improvement that has made all the difference

OTHER OUTCOMES:
Depression severity during screening, and suicidal ideation during treatment | Screening, item 9 weekly up to 9 weeks
  Montgomery Asberg Depression Rating Scale - Self-rated, MADRS-S. Self-rated, range 0 to 60, a higher score indicates higher more depressive symptoms
Alcohol use at screening | Screening
  Alcohol Use Disorders Identification Test. Self-rated, range 0 to 40, a higher score indicates more problematic alcohol use
Drug use at screening | Screening
  Drug Use Disorders Identification Test. Self-rated, range: 0-44. A higher score indicates more problematic substance use
Change in pain-related avoidance behavior over the main phase, as modelled using data from all 11 assessments from pre-treatment assessment, weekly to the primary endpoint (10 weeks). | Pre-treatment, weekly up to 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  The Psychological Inflexibility in Pain Scale-avoidance subscale, PIPS-avoid. Self-rated, range 8-56. A higher score indicates more pain-related avoidance behaviors.
Change in pacing and overdoing behavior over the main phase, as modelled using data from all 11 assessments from pre-treatment assessment, weekly to the primary endpoint (10 weeks). | Pre-treatment, weekly up to 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  Patterns of Activity Measure - Pain, Short form: pacing and overdoing subscales, POAM-P-sf, p/o. Self-rated, range 0-40. A higher score indicates higher degree of pacing and overdoing.
Change in catastrophizing over the main phase, as modelled using data from all 11 assessments from the pre-treatment assessment, weekly to the primary endpoint (10 weeks). | Pre-treatment, weekly up to10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  Pain Catastrophizing Scale, PCS. Self-rated, range 0-52. A higher score indicates a higher degree of pain catastrophizing
Change in hypervigilance over the main phase, as modelled using data from all 11 assessments from pre-treatment assessment, weekly to the primary endpoint (10 weeks). | Pre-treatment, weekly up to 10 weeks. Secondary analyses incorporate 6- and 12-months follow-up assessments.
  Pain Vigilance and Awareness Questionnaire, PVAQ. Self-rated, range 0-80. A higher score indicates more hypervigilance and awareness to pain.
Change in physical activity over the main phase, as modelled using data from all 11 assessments from the pre-treatment assessment, weekly to the primary endpoint (10 weeks). | Pre-treatment, weekly up to 10 weeks.
  The Godin-Shephard leisure-time physical activity questionnaire, GSLTPAQ. Self-rated, range 0-99. A higher score indicates more blocks of at least 15 minutes of physical activity
Treatment credibility and expectancy of improvement at week 3 of main phase | Week 3 of main phase
  Credibility/Expectancy scale (C/E-scale). Self-rated, range: 0-50. A higher score indicates higher credibility/expectancy
Working alliance with therapist at week 3 of main phase | Week 3 of main phase.
  Working alliance inventory-Short, Internet version, WAI-S-Internet. Self-rated, range: 7-144. A higher score indicates better relationship with the therapist.
Client satisfaction with treatment at primary endpoint assessment (10 weeks) | 10 weeks
  Client Satisfaction Questionnaire, CSQ-8. Self-rated, range: 8-32. A higher score indicates higher satisfaction with treatment.
Change in health-related quality of life over the main phase. Data from pre-treatment assessment, the primary endpoint (10 weeks), and the 6- and 12-month follow-up are used for health economic analysis focusing on the main phase | Pre-treatment, 10 weeks, 6- and 12-month follow-up.
  EuroQol 5D, EQ-5D. Self-rated, range: 0-1, i.e., scored as utility for the purpose of calculating quality-adjusted life years for health economic analysis. A higher utility score indicates a higher health-related quality of life
Change in resource use and medications over the main phase. Data from pre-treatment assessment, the primary endpoint, and the 6- and 12-month follow-up are used for health economic analysis focusing on the main phase. | Pre-treatment, 10 weeks, 6- and 12-months follow-up
  Trimbos Institute and Institute of Medical Technology Questionnaire for Costs Associated with Psychiatric Illness, TIC-P. This instrument is scored in terms of resource use for the purpose of calculating societal costs for health economic analysis.
Adverse events at primary endpoint assessment (10 weeks). | 10 weeks
  Adverse events measured using free-text items, primarily reported as the total number of reported events

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hedman-Lagerlöf, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Solna
  - Uppsala University, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hedman-Lagerlof M, Gasslander N, Ahnlund Hoffmann A, Bragesjo M, Etzell A, Ezra S, Frostell E, Hedman-Lagerlof E, Ivert C, Liliequist B, Ljotsson B, Hoppe JM, Palmgren J, Spansk E, Sundstrom F, Sarnholm J, Tzavara G, Buhrman M, Axelsson E. Effect of exposure-based vs traditional cognitive behavior therapy for fibromyalgia: a two-site single-blind randomized controlled trial. Pain. 2024 Jun 1;165(6):1278-1288. doi: 10.1097/j.pain.0000000000003128. Epub 2023 Dec 15. PMID 38131181

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study protocol including rudimentary data analysis plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT05058911/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Detailed information on data analysis (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT05058911/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan for mediation analysis (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT05058911/SAP_002.pdf